CLINICAL TRIAL: NCT02000232
Title: Impact of Unapproved Drug Initiative on Colchicine Use
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: 1U01FD004257-01 (FDA)
Record Dates: First submitted 2013-11-06; First posted 2013-12-04 (Estimated); Last update posted 2022-08-10 (Actual); Status verified 2022-08

CONDITIONS: Gout
Keywords: gout; colchicine
MeSH Terms: conditions — Gout

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Diagnosis with Gout and use of colchicine: Observational study age 18+

SUMMARY:
Measure if FDA regulation of Colchicne in 2009 has resulted in safer use in clinical settings.

Our study will assess the impact of this Initiative on colchicine use and will provide data that supports its continuation and expansion.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of gout
* Current use of colchicine/colcrys to treat gout
* Ablility to provide Informed consent

Exclusion Criteria:

-Inability to provide Informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults diagnosed with gout. Patient's from Stanford hospital and clinics and VA Palo Alto Heath care system are eligible
Sampling Method: Non-Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Frequency of use of colchicine in an unapproved fashion in contemporary medical proactice. | This is an oberservational study and patients will be followed for upto 2 years from enrollment.
  We expect to understand the impact of regulatory approach to colchicine preparation and how marketing can affect clinical use patterns in the real world.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States